CLINICAL TRIAL: NCT04933019
Title: Detection of Clindamycin Resistance Antibiotic Genes Among Staphylococcus Isolates by Using Real Time PCR
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alzahraa Nasser Mahmoud, Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR, Sohag University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-06-14
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Staphylococcus Isolates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clindamycin Resistance Genes among Staphylococcus Isolates by Using Real Time PCR (Other)
  Interventions: Genetic: Detection of Clinclidamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR
- Clindamycin sensetive Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR (Other)
  Interventions: Genetic: Detection of Clinclidamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR

INTERVENTIONS:
Genetic: Detection of Clinclidamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR — Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR

SUMMARY:
Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR

DETAILED DESCRIPTION:
Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR

ELIGIBILITY:
Inclusion Criteria:

* all staphylococcus isolates resistant to clindamycin

Exclusion Criteria:

* non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR | 1 year
  Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Detection of Clindamycin Resistance Antibiotic Genes among Staphylococcus Isolates by Using Real Time PCR